CLINICAL TRIAL: NCT04047316
Title: Development and Validation of a New Digital Dermatoscope in the United States
Status: Completed | Type: Observational
Sponsor: Barco NV (Industry)
Responsible Party: Sponsor
Other Study IDs: CI-PROT-0029
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Digital dermoscopy — Acquire skin images with a new digital dermatoscope

SUMMARY:
A completely new type of digital dermatoscope has been developed in order to take a significant step forward in technology for skin cancer imaging. By means of this study a better insight can be gained of the current performance and workflow in clinical dermatoscopy. This knowledge will be used to further improve the developed technology.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Male or Female, aged less than 18 years, with informed consent of their legally authorized representative.
* Patient presenting with any visible skin lesion for dermatologist review on a body site amenable to optimal photographic imaging.
* Able and willing to comply with all study requirements.
* Patient with a skin lesion that is clinically diagnosed by a dermatologist as benign, malignant or a suspicious skin lesion requiring excisional biopsy for histological diagnosis.

Exclusion Criteria:

* Patients aged under 18 years old where the legally authorized representative is unable or unwilling to provide their informed consent.
* Patients unable to provide informed consent.
* Skin lesions in an anatomical site which is not suitable for photography including hair-obscured site, subungual lesion or inaccessible mucosal site.
* Lesion is at a site where previous surgery was undertaken.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be considered for enrollment in the study when they have a lesion that is accessible to the new digital dermatoscope and are able to give informed consent (guardian in case of patients under 18 years).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Performance of the new device in its normal conditions of use | 6 months
  The outcome will be measured by a questionnaire with performance-related questions for clinicians to answer about a set of images from the collected database. A Likert-based scale will be used for the answers: from highly agree to highly disagree.
Usability of the new device | 1 month
  The outcome will be measured by a questionnaire with usability-related questions for clinicians.
Safety of the new device in its normal conditions of use | 1 year
  The number of adverse events will be reported to assess safety of the device.

SECONDARY OUTCOMES:
Develop a database of skin images with the new device with metadata and histopathology of excised lesions | 1 year
  The outcome of the secondary objective will be an anonymized database of digital skin lesion images and corresponding metadata and a set of high quality images amenable to clinician evaluation.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dermatologic Surgery Center of Washington LLC, Chevy Chase, Maryland
  - Silver Falls Dermatology, Salem, Oregon